CLINICAL TRIAL: NCT01902342
Title: A Clinical Trial to Investigate the Influence of CES1 Polymorphism on Pharmacokinetic Characteristics of Oseltamivir in Healthy Korean Volunteers
Brief Title: A Clinical Trial to Investigate the Influence of CES1 Polymorphism on Oseltamivir
Acronym: CES1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CES01
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CES1 gene variant group (Experimental): Oseltamivir 75 mg 1 cap
  Interventions: Drug: Oseltamivir 75 mg 1 cap
- CES1 gene wild type group (Experimental): Oseltamivir 75 mg 1 cap
  Interventions: Drug: Oseltamivir 75 mg 1 cap

INTERVENTIONS:
Drug: Oseltamivir 75 mg 1 cap
  Other Names: Tamiflu

SUMMARY:
Investigate genetic variability of CES1 gene on pharmacokinetics of oseltamivir in healthy Korean volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

1. Agreement with written informed consent
2. Adult healthy male or female subject age 20 to 45

Exclusion Criteria:

1. Clinically significant, active gastrointestinal system, cardiovascular system, pulmonary system, renal system, endocrine system, blood system, digestive system, central nervous system, mental disease or malignancy
2. Medication with any drug which may affect the pharmacokinetics of oseltamivir within 14 days
3. Previously donate whole blood within 30 days or Previously participated in other trial within 60 days
4. Subject with known for hypersensitivity reactions to oseltamivir
5. Subject who perform contraception during study periods
6. Female woman who are pregnant or are breast feeding
7. An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Oseltamivir pharmacokinetic parameters | Up to 0 to 48 h post dose
  Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast and AUCinf)
Oseltamivir carboxylate pharmacokinetic parameters | Up to 0 to 48 h post dose
  Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast and AUCinf)

SECONDARY OUTCOMES:
Other oseltamivir pharmacokinetic parameters | Up to 0 to 48 h post dose
  first time to reach Cmax (tmax), terminal half-life (t1/2z), apparent clearance (CL/F), apparent renal clearance (CLR/F), metabolic ratio
Other oseltamivir carboxylate pharmacokinetic parameters | Up to 0 to 48 h post dose
  first time to reach Cmax (tmax), terminal half-life (t1/2z), apparent clearance (CL/F), apparent renal clearance (CLR/F), metabolic ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Soo Lim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

REFERENCES:
- [Derived] Oh J, Lee S, Lee H, Cho JY, Yoon SH, Jang IJ, Yu KS, Lim KS. The novel carboxylesterase 1 variant c.662A>G may decrease the bioactivation of oseltamivir in humans. PLoS One. 2017 Apr 24;12(4):e0176320. doi: 10.1371/journal.pone.0176320. eCollection 2017. PMID 28437488